CLINICAL TRIAL: NCT07260084
Title: Prognostic Impact of Frailty in Cardiogenic Shock: Nationwide Cohort Study
Brief Title: Prognostic Impact of Frailty in Cardiogenic Shock
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ki Hong Choi, Professor, Samsung Medical Center
Other Study IDs: CS Frailty
Record Dates: First submitted 2025-09-24; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Cardiogenic Shock; Frailty; Age
Keywords: frailty; cardiogenic shock; Hospital Frailty Risk Score; Age
MeSH Terms: conditions — Shock, Cardiogenic; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to show prognostic impact of frailty in cardiogenic shock according to age. The main questions it aims to answer are:

* Can frailty successfully predict outcomes in cardiogenic shock?
* Whether the impact of frailty would differ with age in cardiogenic shock?

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years who were admitted to the intensive care unit (ICU) of tertiary hospitals and were diagnosed with CS

Exclusion Criteria:

* Patients diagnosed with anaphylaxis
* Patients with a documented history of shock in the year before the index admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged ≥18 years who were admitted to the intensive care unit (ICU) of tertiary hospitals and were diagnosed with CS
Sampling Method: Non-Probability Sample
Enrollment: 207419 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
In-hospital all-cause mortality | During index hospitalization for cardiogenic shock (up to hospital discharge)
  Death from any cause occurring during the index hospitalization for cardiogenic shock. Number of participants with the event was measured

SECONDARY OUTCOMES:
Heart failure-related rehospitalization | From index hospitalization until 15 years of follow-up.
  Any inpatient admission with a primary or secondary diagnosis of heart failure (ICD-10 I50.x), identified from claims data and prescription records.Number of participants with the event was measured.
Cognitive impairment | From index hospitalization until 15 years of follow-up.
  New-onset cognitive dysfunction after discharge, defined using ICD-10 codes (R41.x for memory disturbance, F06.7 for mild cognitive disorder) or new diagnosis of dementia (F00-F03, G30) or prescription of anti-dementia medications (donepezil, rivastigmine, galantamine, memantine). Number of participants with event was measured
Mental health problems | From index hospitalization until 15 years of follow-up.
  Composite of new-onset psychiatric diagnoses after discharge including 6 domains defined using ICD-10 codes. Domains include depression (ICD-10 F32-F33), anxiety disorders (F41.x), somatization disorder (F45.x), stress-related disorders (F43.x), sleep disorders (G47.x), and substance use disorders (F10-F19). Diagnostic codes supported by prescription data (e.g., antidepressants, anxiolytics). Number of participants with the event was measured.
Long-term all-cause mortality | From index hospitalization until 15 years of follow-up.
  Death from any cause, identified with the Statistics Korea nationwide death registry. Number of participants with the event was measured.